CLINICAL TRIAL: NCT04308434
Title: CSD190601: A Study to Determine Subject Puffing Patterns of Electronic Nicotine Delivery Systems in an Ambulatory Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD190601
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- CSD190601-11 (Experimental): Subjects will self-assign to flavor variant CSD190601-11 of 1.5% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-11
- CSD190601-12 (Experimental): Subjects will self-assign to flavor variant CSD190601-12 of 1.5% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-12
- CSD190601-13 (Experimental): Subjects will self-assign to flavor variant CSD190601-13 of 1.5% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-13
- CSD190601-14 (Experimental): Subjects will self-assign to flavor variant CSD190601-14 of 1.5% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-14
- CSD190601-15 (Experimental): Subjects will self-assign to flavor variant CSD190601-15 of 1.5% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-15
- CSD190601-16 (Experimental): Subjects will self-assign to flavor variant CSD190601-16 of 1.5% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-16
- CSD190601-17 (Experimental): Subjects will self-assign to flavor variant CSD190601-17 of 1.5% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-17
- CSD190601-21 (Experimental): Subjects will self-assign to flavor variant CSD190601-21 of 3.0% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-21
- CSD190601-22 (Experimental): Subjects will self-assign to flavor variant CSD190601-22 of 3.0% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-22
- CSD190601-23 (Experimental): Subjects will self-assign to flavor variant CSD190601-23 of 3.0% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-23
- CSD190601-24 (Experimental): Subjects will self-assign to flavor variant CSD190601-24 of 3.0% ENDS products based on their preferred flavor.,
  Interventions: Other: CSD190601-24
- CSD190601-25 (Experimental): Subjects will self-assign to flavor variant CSD190601-25 of 3.0% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-25
- CSD190601-26 (Experimental): Subjects will self-assign to flavor variant CSD190601-26 of 3.0% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-26
- CSD190601-27 (Experimental): Subjects will self-assign to flavor variant CSD190601-27 of 3.0% ENDS products based on their preferred flavor.
  Interventions: Other: CSD190601-27

INTERVENTIONS:
Other: CSD190601-11 — Flavor variant CSD190601-11 of a 1.5% nicotine ENDS product
  Arms: CSD190601-11
Other: CSD190601-12 — Flavor variant CSD190601-12 of a 1.5% nicotine ENDS product
  Arms: CSD190601-12
Other: CSD190601-13 — Flavor variant CSD190601-13 of a 1.5% nicotine ENDS product
  Arms: CSD190601-13
Other: CSD190601-14 — Flavor variant CSD190601-14 of a 1.5% nicotine ENDS product
  Arms: CSD190601-14
Other: CSD190601-15 — Flavor variant CSD190601-15 of a 1.5% nicotine ENDS product
  Arms: CSD190601-15
Other: CSD190601-16 — Flavor variant CSD190601-16 of a 1.5% nicotine ENDS product
  Arms: CSD190601-16
Other: CSD190601-17 — Flavor variant CSD190601-17 of a 1.5% nicotine ENDS product
  Arms: CSD190601-17
Other: CSD190601-21 — Flavor variant CSD190601-21 of a 3.0% nicotine ENDS product
  Arms: CSD190601-21
Other: CSD190601-22 — Flavor variant CSD190601-22 of a 3.0% nicotine ENDS product
  Arms: CSD190601-22
Other: CSD190601-23 — Flavor variant CSD190601-23 of a 3.0% nicotine ENDS product
  Arms: CSD190601-23
Other: CSD190601-24 — Flavor variant CSD190601-24 of a 3.0% nicotine ENDS product
  Arms: CSD190601-24
Other: CSD190601-25 — Flavor variant CSD190601-25 of a 3.0% nicotine ENDS product
  Arms: CSD190601-25
Other: CSD190601-26 — Flavor variant CSD190601-26 of a 3.0% nicotine ENDS product
  Arms: CSD190601-26
Other: CSD190601-27 — Flavor variant CSD190601-27 of a 3.0% nicotine ENDS product
  Arms: CSD190601-27

SUMMARY:
This study will be a single-center, controlled, open-label, parallel two-study-group investigation to evaluate the puffing patterns of healthy adult consumers of tobacco products switching from a usual brand (UB) Electronic Nicotine Delivery Systems (ENDS) product to one of two different ENDS, Product A with 1.5% nicotine, and Product B with 3.0% nicotine, over a three-week ambulatory period. This study will be conducted in support of a Premarket Tobacco Product Application (PMTA) ENDS submission to the US Food and Drug Administration (FDA) Center for Tobacco Products (CTP).

DETAILED DESCRIPTION:
Potential subjects may complete a pre-screening interview (by phone) and will complete a Screening Visit to assess their eligibility. Based on meeting eligibility requirements, it is desirable that subjects will be enrolled into the study on the same day of their Screening Visit. However, because of delays in receiving clinical laboratory test results, additional time may be needed to complete Enrollment. It may be necessary that subjects will need to return to the clinic on another day to compete Enrollment.

To minimize bias, subjects will be assigned to either Product A or Product B based on the scheduled visit to the clinic during Screening and Enrollment. Subjects will then be assigned to one of the seven e-liquid flavor variants for either Product A or Product B. Subjects will be allowed to sample or try flavors and determine which flavor that they would like to use for the length of the study.

At the Screening/Enrollment visit, subjects will be provided an orientation to the product, including the power unit and cartridges for their assigned product, and the corresponding Product Use and Behavior (PUB) instrument, PUB application, and an electronic device provided by the Sponsor. Based upon their UB ENDS usage, they will be given a sufficient amount (for three weeks of ad libitum use equaling 375% of their self-reported UB reported weekly use) of their assigned Product A or Product B cartridges.

The study will involve a one-week acclimation period followed by a two-week product use evaluation period. Subjects will be instructed to use their assigned Product A or Product B product in place of their UB ENDS during the three-week study period, but they will be allowed to use non-ENDS tobacco/nicotine-containing products according to their normal use pattern. The PUB instrument will collect topography data, and product use data will be uploaded frequently using a web-based PUB application installed on the electronic device provided by the Sponsor.

At the end of the first week of the study, subjects will receive a phone call from the clinic to assess Investigational Product (IP) compliance and to ensure that they are not using their UB ENDS. Throughout the study, subjects will receive weekly phone calls at a minimum to remind them of guidelines for using their assigned IP. All used cartridges may be disposed of by the subject.

At the conclusion of the three-week ambulatory period, the subjects will return to the clinic, return the Product A or Product B power unit, any associated USB charger, all unused IP cartridges, the corresponding PUB instrument and its charger, and the provided electronic device. Each subject will complete all End of Study procedures including completing the Product Evaluation Scale (PES) questionnaire, and then subjects will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female, ≥ 21 years of age, inclusive, at the time of consent.
3. Positive urine cotinine test at Screening.
4. Cartridge-based, closed-system ENDS are the primary form of tobacco/nicotine-containing products used within 30 days of Screening. Subjects may be users of other tobacco/nicotine-containing products. If the subject is a dual/poly user of tobacco/nicotine-containing products then the subject must self report that a cartridge-based, closed-system ENDS is their primary product.
5. Must have used 2 or more cartridges per week over the last 30 days. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the Principal Investigator (PI).
6. Females must be willing to use a form of contraception acceptable to the PI from the time of signing the ICF until the end of the study.
7. Must be willing to use the assigned IP and only the assigned flavor as their exclusive source of ENDS use for the full duration of the three-week ambulatory period. Use of other non-ENDS tobacco/nicotine-containing products will be permitted during the ambulatory period.
8. Must have familiarity with modern electronic devices such as an IOS/Android smart phone or tablet computer ("tablet") and be willing to be provided an electronic device, that allows for both Bluetooth connectivity and internet connectivity and be willing to keep both active for the length of the study.
9. Must be willing to use an application on the provided electronic device, and keep the application active for the length of the study.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study participant unsuitable to participate in this clinical study.
2. History or presence of diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes, with exceptions at the PI's discretion.
4. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening-Enrollment Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
6. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (NRT, e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
7. Participation in another clinical trial within (≤) 30 days prior to signing the ICF. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
8. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
9. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
10. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening.
11. Postpones a decision to quit using tobacco/ nicotine-containing products in order to participate in this study or a previous attempt within (≤) 30 days prior to the signing of the ICF.
12. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol breathalyzer result at Screening.
13. Determined by the PI to be inappropriate for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Arithmetic Mean | 2 weeks
  Arithmetic Mean puff duration

CONTACTS AND LOCATIONS:
Overall Officials: Gary Dull, PhD, Study Director — RAIS
Locations (1):
- Clinical Research Atlanta, Stockbridge, Georgia, United States

IPD SHARING:
Plan to Share IPD: No